CLINICAL TRIAL: NCT00088608
Title: A Multicenter, Open Label Study to Assess the Safety and Efficacy of 600 µg SOM230, Administered Subcutaneously, b.i.d. in Patients With Cushing's Disease
Brief Title: A Study to Assess SOM230 in Patients With Pituitary Cushing's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2208
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Cushing's Syndrome
MeSH Terms: conditions — Cushing Syndrome

INTERVENTIONS:
Drug: SOM230 s.c.

SUMMARY:
The study treatment period is 15 days in length and includes patients with pituitary Cushing's disease who are candidates for surgical intervention as well as and patients who have recurrent Cushing's post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pituitary Cushing's disease within the two months prior to study entry
* Patients for whom written informed consent to participate in the study has been obtained
* Female patients of child bearing potential who have not undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation must agree to use barrier contraception throughout the course of the study, and for one month after the study has ended

Exclusion Criteria:

* Female patients who are pregnant or lactating
* Patients who have been previously treated with certain medications may be required to be without certain medications prior to entering the study
* Poorly controlled diabetes mellitus as indicated by the presence of ketoacidosis or HgbA1C > 10
* Patients who have congestive heart failure, unstable angina, cardiac arrhythmia or history of acute MI less than one year prior to the study entry or clinically significant impairment in cardiovascular function (e.g. blood pressure of 190/100mmHg or greater)
* Patients with chronic liver disease
* Patients with clotting disorders or abnormal blood counts
* History of immuno-compromise, including a positive HIV test result
* Patients with active gall bladder disease
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Patients with active malignant disease (with the exception of basal cell carcinoma or carcinoma in situ of the cervix)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-04; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Urinary Free Cortisol after 15 days of treatment

SECONDARY OUTCOMES:
Serum cortisol
ACTH
Clinical manifestations
Pharmacokinetics
Safety
Tolerability
Development of biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Cedars-Sinai Pituitary Center, Los Angeles, California
  - Massachusetts General Hospital NE Unit, Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Midwest Endocrinology Associates, Milwaukee, Wisconsin

REFERENCES:
- [Result] Boscaro M, Ludlam WH, Atkinson B, Glusman JE, Petersenn S, Reincke M, Snyder P, Tabarin A, Biller BM, Findling J, Melmed S, Darby CH, Hu K, Wang Y, Freda PU, Grossman AB, Frohman LA, Bertherat J. Treatment of pituitary-dependent Cushing's disease with the multireceptor ligand somatostatin analog pasireotide (SOM230): a multicenter, phase II trial. J Clin Endocrinol Metab. 2009 Jan;94(1):115-22. doi: 10.1210/jc.2008-1008. Epub 2008 Oct 28. PMID 18957506
- [Derived] Trementino L, Cardinaletti M, Concettoni C, Marcelli G, Polenta B, Spinello M, Boscaro M, Arnaldi G. Salivary cortisol is a useful tool to assess the early response to pasireotide in patients with Cushing's disease. Pituitary. 2015 Feb;18(1):60-7. doi: 10.1007/s11102-014-0557-x. PMID 24482099